CLINICAL TRIAL: NCT05931458
Title: ADVANCED-UC TRIAL: AppenDectomy Vs ANti TNF-a in Inducing Clinical and EnDoscopic Remission in Left-sided Ulcerative Colitis - A Randomized Clinical Trial
Brief Title: AppenDectomy Vs ANti TNF-a in Inducing Clinical and EnDoscopic Remission in Left-sided Ulcerative Colitis
Acronym: ADVANCED-UC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Gaetano Luglio, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 340/21
Record Dates: First submitted 2023-06-18; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Appendectomy; Infliximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Infliximab
  Interventions: Drug: Infliximab
- Group 2 (Experimental): Appendectomy
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Laparoscopic appendectomy is a relatively simple surgical procedure that can be performedby most surgeons, either on an outpatient basis or with a single-night hospital stay. The laparoscopic approach is now the recommended option due to faster recovery times and fewer wound complications.
  Arms: Group 2
Drug: Infliximab — Administration of Infliximab (Anti-TNF-a biologic drug)
  Arms: Group 1

SUMMARY:
Ulcerative Colitis (UC) is a chronic Inflammatory Bowel Disease (IBD) characterized by a multifactorial etiology, a variable involvement of large bowel, and a relapsing-remitting course.

In order to keep the disease in a "quiescent" status and to prevent relapses, a significative percentage of UC patients will remain on long-term drug therapy. However, long-term immunosuppressant therapy is not free of risks and complications: in fact, these therapies have an impact on both healthcare system resources and patients' quality of life; more, there are even concerns regarding the side effects of long-term immunosuppressant therapy.

Over the past 20 years, a considerable amount of evidence was produced to support the immunomodulatory role of the appendix in the development and course of UC: there is a strong inverse relationship between previous appendectomy and development of the UC. One of the proposed theories to justify this link is that the appendix could act as a reservoir for commensal bacteria that can be secreted into the colon, affecting its microbiome and immunological response; another theory describes the appendix as the "priming site" for the cytokine production and the immunological cascade that may trigger inflammation in colon and rectum.

The idea of this study moves from these assumptions: the investigators aim to evaluate the impact of appendectomy in patients with UC who are candidates to the treatment with biologics (Anti TNF-a), because of conventional therapies failure. To further reduce any ethical problems and significantly lower any surgical morbidity, investigators will restrict the study population to only patients with active left-sided colitis, so that the surgery for appendectomy will take place on a non-inflamed cecum.

By undertaking this study, the investigators hope to a) learn more about the role of appendix and the impact of appendectomy in the clinical history of Ulcerative Colitis; b) demonstrate that laparoscopic appendectomy, a relatively simple surgical procedure that can also be performed in day-surgery with a very low expected complication rate, is a treatment that is superior to biological therapy, avoiding patients starting a chronic, long-lasting therapy, with the consequent risk of immunosuppression, and with possible higher costs for the health system in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or above
* Patients with a confirmed diagnosis of left-sided UC (extended up to the mid transverse colon)
* Patients with active disease refractory to conventional treatment and candidates for anti- TNF-a treatment
* Patients who have given consent to the surgical procedure

Exclusion Criteria:

* Patients under the age of 18
* Lack of diagnostic certainty of Ulcerative Colitis / Crohn's disease diagnostic doubt
* Patients who previously received appendectomy
* Patients who have had previous laparotomic abdominal surgery, which could make the appendectomy more complex
* Patients with Severe Acute Colitis/Toxic Megacolon
* Patients who have not given their consent to the intervention
* Patients who receive a different surgical procedure from appendectomy because of intraoperative complications
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Steroid Free Clinical Remission | 3 months
  Steroid Free Clinical Remission at 3 and 12 months (defined as Partial Mayo score </=2, with no individual sub-score >1)
Steroid Free Clinical Remission | 12 months
  Steroid Free Clinical Remission at 3 and 12 months (defined as Partial Mayo score </=2, with no individual sub-score >1)
Endoscopic remission | 3 months
  Endoscopic remission at 3 and 12 months (defined as MAYO CU score </ = 1)
Endoscopic remission | 12 months
  Endoscopic remission at 3 and 12 months (defined as MAYO CU score </ = 1)
Assessment of Quality of Life | 3 months
  Assessment of Quality of Life at 3 and 12 months, through the SIBDQ (Short Inflammatory Bowel Disease Questionnaire, ranging from 10, meaning poor quality of life, to 70, meaning optimal quality of life)
Assessment of Quality of Life | 12 months
  Assessment of Quality of Life at 3 and 12 months, through the SIBDQ (Short Inflammatory Bowel Disease Questionnaire, ranging from 10, meaning poor quality of life, to 70, meaning optimal quality of life)
Assessment of Quality of Life | 3 months
  Assessment of Quality of Life at 3 and 12 months, through the SF-36 questionnaire (Short-form 36)
Assessment of Quality of Life | 12 months
  Assessment of Quality of Life at 3 and 12 months, through the SF-36 questionnaire (Short-form 36)

SECONDARY OUTCOMES:
Clinical Response | 3 months
  Clinical Response at 3 and 12 months (defined as a reduction of the MAYO SCORE of at least 3points). MAYO SCORE ranges from 0 (inactive disease) to 3 (severe disease activity).
Clinical Response | 12 months
  Clinical Response at 3 and 12 months (defined as a reduction of the MAYO SCORE of at least 3points). MAYO SCORE ranges from 0 (inactive disease) to 3 (severe disease activity).
Failure rate | 3 months
  Evaluation of the failure rate at 3, 12 and 24 months (evaluated as the rate of use of the biological or colectomy in the "treatment" group, as the rate of use of a second biological or colectomy in the "control" group)
Failure rate | 12 months
  Evaluation of the failure rate at 3, 12 and 24 months (evaluated as the rate of use of the biological or colectomy in the "treatment" group, as the rate of use of a second biological or colectomy in the "control" group)
Failure rate | 24 months
  Evaluation of the failure rate at 3, 12 and 24 months (evaluated as the rate of use of the biological or colectomy in the "treatment" group, as the rate of use of a second biological or colectomy in the "control" group)
Complication assessment | 30 days
  Complication assessment: Treatment-related serious adverse events will be compared between the two groups. The Dindo-Clavien Classification will be used within 30 days of the procedure in patientsundergoing appendectomy. For patients undergoing biologics, the cumulative rate of treatment- related serious adverse events up to 12 months will be considered. Hospitalization rates will also be assessed as a consequence of adverse events to treatment.
Complication assessment | 12 months
  Complication assessment: Treatment-related serious adverse events will be compared between the two groups. The Dindo-Clavien Classification will be used within 30 days of the procedure in patientsundergoing appendectomy. For patients undergoing biologics, the cumulative rate of treatment- related serious adverse events up to 12 months will be considered. Hospitalization rates will also be assessed as a consequence of adverse events to treatment.
Histological remission | 3 months
  Evaluation of histological remission at 3 and 12 months with the Geboes score (ranging from 0, histological remission, to 22, severe inflammatory injury).
  In patients undergoing appendectomy, the appendix will also be histologically evaluated with the same Geboes score in addition to the presence of PARP (peri-appendicular patches).
Histological remission | 12 months
  Evaluation of histological remission at 3 and 12 months with the Geboes score (ranging from 0, histological remission, to 22, severe inflammatory injury).
  In patients undergoing appendectomy, the appendix will also be histologically evaluated with the same Geboes score in addition to the presence of PARP (peri-appendicular patches).
Immunohistochemical evaluation | 3 months
  Immunohistochemical evaluation of the IgA / IgG ratio and correlation between the findings onthe appendix and the findings on colonic biopsy at 3 and 12 months.
Immunohistochemical evaluation | 12 months
  Immunohistochemical evaluation of the IgA / IgG ratio and correlation between the findings onthe appendix and the findings on colonic biopsy at 3 and 12 months.
Colectomy rate | 12 months
  Evaluation of "Colectomy rate" at 12, 24 and 60 months
Colectomy rate | 24 months
  Evaluation of "Colectomy rate" at 12, 24 and 60 months
Colectomy rate | 60 months
  Evaluation of "Colectomy rate" at 12, 24 and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Luglio, Prof, Principal Investigator — Federico II University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After the end of the study